CLINICAL TRIAL: NCT05758545
Title: Concurrent Optical and Magnetic Stimulation (COMS) for Treatment of Refractory Diabetic Foot Ulcer; a Prospective Randomized, Sham-controlled, Double-blinded, Pivotal Clinical Trial
Brief Title: Trial to Evaluate the Safety and Effectiveness of Treatment With COMS One Device in Subjects With Diabetic Foot Ulcers
Acronym: Mavericks
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Piomic Medical (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COMS_03
Record Dates: First submitted 2023-02-09; First posted 2023-03-07 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-09

CONDITIONS: Diabetic Foot Ulcer
Keywords: Refractory Diabetic Foot Ulcer (DFU)
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: The purpose of this clinical trial is to evaluate the safety and effectiveness of the treatment with the COMS One device in subjects with refractory diabetic foot ulcers (DFUs). The prospective randomized, double-blinded, sham-controlled trial is designed to demonstrate superiority of wound closure of the COMS One device to a sham-control device through 24 weeks post-application, when each is administered in conjunction with standard of care (SOC) in the treatment of DFUs.
  Following randomization, subjects will be assigned treatment with either COMS One device or the Sham device in conjunction with SOC. At least 50% of subjects are required to be 65 years or older at randomization.
  Prospective, randomized, double-blinded, placebo-controlled trials provide the most objective methods for analyzing the outcomes of multiple treatment groups. The blinded use of a sham device allows for a true comparison of COMS One treatment in conjunction with SOC to SOC alone.
Who Masked: Participant, Investigator
Masking Description: Permuted block randomization will be applied to generate randomization codes using a mix of blocks of size 2 and 4. Randomization will be stratified by site and age (<65 years, ≥65 years). Both the COMS One device and the Sham device will be prepared to appear to be identical to the subject to achieve the double-blind purposes and each device will be given a unique serial identifier.
  To avoid assessment bias, each site will have an Inter-observer (blinded assessor) who will be blinded to treatment and perform and document all assessments of the target DFU evolution. Following target DFU assessment, the treatment will be performed by another assigned clinician, who will not have any involvement with the Inter-observer. Furthermore, both parties will be instructed not to discuss target DFU evolution or treatment with each other. This will provide an adequate level of masking to ensure that the trial is double-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- COMS One device (Active Comparator): The COMS One device is the housing unit for the user controls, displays and functions including embedded software, lithium-ion battery, optical (LEDs) and a magnetic stimulation coil. The COMS One device is reusable (the component can be used on multiple subjects and is cleaned between uses).
  The COMStouch is a sterile single-use component. The COMStouch provides a base and sterile barrier for the COMS One device.
  The COMSfix component is a self-adhesive single-use strap used to hold the COMS One device and COMStouch components in place during treatment.
  Interventions: Device: COMS One device
- Sham device (Sham Comparator): The sham device is the housing unit for the user controls, displays and functions including embedded software, lithium-ion battery, optical (LEDs) and a magnetic stimulation coil. The sham device is reusable (the component can be used on multiple subjects and is cleaned between uses).
  The COMStouch is a sterile single-use component. The COMStouch provides a base and sterile barrier for the sham device.
  The COMSfix component is a self-adhesive single-use strap used to hold the sham device and COMStouch components in place during treatment.
  Interventions: Device: Sham device

INTERVENTIONS:
Device: COMS One device — The COMS One device incorporates technologies for optical and magnetic stimulation. The optical stimulation component is designed to emit light by two types of light emitting diodes (LEDs) in the wavelength of 660 nm (red) and 830 nm (near infrared) range of the electromagnetic spectra. The magnetic stimulation component is generated by a coil emitting pulse modulated magnetic fields in the extremely low frequency (ELF) range of the electromagnetic spectra. The COMS One is a lightweight, portable device. The device is locally applied via a single use disposable component (COMStouch) that provides a base and sterile barrier for the unit. The device is attached via a single use strap (COMSfix). The device has been slightly adapted in order to make sure blinding is achieved/maintained. The specific feature that has been modified for the purpose of blinding is sensor detecting whether the device is lying on the skin.
  Other Names: Concurrent Optical and Magnetic Stimulation
  Arms: COMS One device
Device: Sham device — The Sham device is a lightweight, portable device. The device is applied via a single use disposable component (COMStouch) that provides a base and sterile barrier for the unit. The device is attached via a single use strap (COMSfix). The device has been slightly adapted in order to make sure blinding is achieved/maintained. The specific features that have been modified for the purposes of blinding include the following: 1) therapeutic output, and 2) sensor detecting whether the device is lying on the skin.
  Arms: Sham device

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and effectiveness of the treatment with the COMS One device in subjects with refractory diabetic foot ulcers (DFUs). The prospective randomized, double-blinded, sham-controlled trial is designed to demonstrate superiority of wound closure of the COMS One device to a sham-control device through 24 weeks post-application, when each is administered in conjunction with standard of care (SOC) in the treatment of DFUs.

DETAILED DESCRIPTION:
The purpose of this clinical trial is to evaluate the safety and effectiveness of the treatment with the COMS One device in subjects with refractory diabetic foot ulcers (DFUs). The prospective randomized, double-blinded, sham-controlled trial is designed to demonstrate superiority of wound closure of the COMS One device to a sham-control device through 24 weeks post-application, when each is administered in conjunction with standard of care (SOC) in the treatment of DFUs.

Primary Objective:

The COMS One Therapy System is intended to promote wound healing in chronic DFUs. As part of the clinical investigation, the primary objective is to determine time to complete wound healing, defined as complete skin re-epithelialization without drainage confirmed by 2 consecutive trial visits 2 weeks apart.

Secondary Objectives:

Secondary objectives are confirmation of safety and assessment of wound healing parameters as well as subject and site reported outcomes.

A total of 450 subjects with refractory DFU will be screened. It is expected that 50% of subjects will be excluded from the trial if either of the following occurs between screening and randomization: >30% wound closure over a period of 2 weeks or >50% wound closure over a period of 4 weeks (measured post-debridement). The remaining 224 subjects will be randomized into two groups (112 Subjects Sham device treated; 112 Subjects COMS One device treated) to account for approximately 10% missing data due to early trial withdrawal or missed endpoint assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are male or female, ≥22 and ≤90 years of age
2. Female subjects of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers, or abstinence) starting at screening and throughout the duration of their study participation.
3. The participant (or LAR if applicable) must be able to understand and sign the informed consent form (ICF) and comply with requirements set in the protocol including trial visits, trial treatment and dressing regimens and compliance with required offloading device (if applicable)
4. Type 1 or Type 2 diabetes mellitus
5. Presence of one full-thickness DFU located at or below the malleoli (If the subject has more than one DFU that meets eligibility criteria, the investigator will designate one DFU as the target DFU to be treated in the trial)
6. Wagner Grade 1 or 2 (without bone exposure)
7. There is a minimum 2 cm margin between the target DFU and any other ulcer on that same foot, post-debridement
8. Target DFU duration >30 days and <52 weeks
9. Target DFU area between 0.5 - 25 cm2 at screening (Target DFU is ≥ 0.5cm2 after debridement at start of Run-In Phase)
10. Adequate vascular perfusion of the target limb (same limb as where the target DFU is located) as evidenced by: either a skin perfusion pressure (SPP) measurement of ≥30mmHg OR an ankle-brachial index (ABI) >0.7 but less than 1.2 or a toe-brachial index (TBI) >0.4 but less than 1.1 or a transcutaneous oxygen pressure (TcPO2) >40mmHg

Exclusion Criteria:

1. Known pregnancy or lactating
2. Active skin cancer, a history of skin cancer or any other localized cancer, precancerous lesions or large moles in the areas to be treated.
3. Subject who is taking any medications the Investigator believes may interfere with healing of the target DFU
4. Subject who is currently undergoing treatment for an active systemic infection, including osteomyelitis
5. Wagner Grade 3, 4 or 5
6. Participation in another trial with investigational drug or device within the 30 days preceding and during the present trial
7. Any co-morbid medical condition which places the subject at unreasonable risks in the opinion of the Investigator
8. Subject has chronic renal insufficiency requiring dialysis (end stage renal disease)
9. Subject is being treated with systemic corticosteroids (prednisone, dexamethasone, hydrocortisone, methylprednisolone, or similar) >10mg/day for more than 10 days or any dose >30 days
10. For subjects in the 2-Week Run-In Phase: more than 30% closure of target DFU at Screening Run-In Phase Visit I or Randomization/Baseline Visit or more than 50% closure of target DFU between the 2 Week Historical Period and Randomization/Baseline Visit (measured post-debridement)
11. For subjects in the 4-Week Run-In Phase: more than 30% closure of target DFU at Screening Run-In Visit II or between Screening Run-In Phase Visit II and Randomization/Baseline Visit or more than 50% closure of target DFU between Screening Run-In Phase Visit I and Randomization/Baseline Visit (measured post-debridement)
12. Blood chemistry or counts values as follows (based on subject's medical files):

    1. Pre-albumin <10 mg/dL OR albumin <2.8 g/dL
    2. Serum BUN >60 mg/dL
    3. Serum creatinine >4.0 mg/dL
    4. WBC <2.0 x 109/L
    5. Hemoglobin <8.0 g/dL
    6. Absolute neutrophil <1.0 x 109/L
    7. Platelet count <50 x 109/L
    8. HbA1C >12%

Ages: 22 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2027-06-19 (Estimated); Study Completion 2027-06-19 (Estimated)

PRIMARY OUTCOMES:
Complete wound healing | 24 weeks post-application
  The primary endpoint for this pivotal trial is time to complete wound closure from randomization through 24 weeks, which is defined as complete skin re-epithelialization without drainage confirmed by 2 consecutive trial visits 2 weeks apart.

SECONDARY OUTCOMES:
Time to ≥50% wound area reduction | Through 24 weeks
  Time in number of days until wound area is reduced by ≥50% compared to wound area at time of randomization
Time to ≥90% wound area reduction | Through 24 weeks
  Time in number of days until wound area is reduced by ≥90% compared to wound area at time of randomization
Incidence of complete wound closure | 8 week, 12 week, 16 week, 20 week and 24 week
  Incidence of complete wound closure after 8, 12, 16, 20, and 24 weeks, which is defined as complete skin re-epithelialization without drainage
Partial wound closure | 8 week, 12 week, 16 week, 20 week and 24 week
  Percent Wound Area Reduction (PWAR) at week 8, 12, 16, 20, 24
Incidence of all related or serious adverse events | Up to week 12 and week 24
  Number of subjects with one or more related adverse event or serious adverse events. Related adverse events are those judged by the investigator to be possibly, probably, or definitely related to the COMS One device or other trial procedures.
Time to target diabetic foot ulcer re-occurrence | Up to 24 weeks
  Time in number of days from randomization until re-occurrence of the target diabetic foot ulcer, assessed up to 24 weeks
Time to amputation | Up to 24 weeks
  Time in number of days from randomization until amputation associated with the target diabetic foot ulcer, assessed up to 24 weeks
Pain assessment | Week 1, Week 8, Week 12, Week 24
  Wong-Baker FACES Pain Rating Scale - patient chooses the face that best demonstrates the physical pain they are experiencing at four time points throughout study participation
Quality of life survey | Week 1, Week 8, Week 12, Week 24
  36-Item Short Form Survey (SF-36) - health-related quality of life questionnaire that is completed by patients at four time points throughout study participation

CONTACTS AND LOCATIONS:
Overall Officials: Aksone Nouvong, DPM, Principal Investigator — University of California, Los Angeles
Locations (26):
- United States (26):
  - Titan Clinical Research, Mesa, Arizona
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - Center for Clinical Research Inc., Castro Valley, California
  - Limb Preservation Platform, Inc., Fresno, California
  - Angel City Research, Inc., Los Angeles, California
  - UCLA Ronald Regan - Department of Surgery, Los Angeles, California
  - Center for Clinical Research Inc., San Francisco, California
  - ILD Research Center, Vista, California
  - Bay Pines VA Healthcare System, Bay Pines, Florida
  - University of Florida Health Jacksonville, Jacksonville, Florida
  - Clever Medical Research LLC, Miami, Florida
  - The Angel Medical Research Corporation, Miami Lakes, Florida
  - Aiyan Diabetes Center, Augusta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Rush University, Chicago, Illinois
  - Gateway Clinical Trials, O'Fallon, Illinois
  - Curalta Clinical Trials, Westwood, New Jersey
  - Veteran Affairs of WNY Healthcare System, Buffalo, New York
  - Northwell Comprehensive Wound Healing Center, Lake Success, New York
  - UNC Medical Center, Chapel Hill, North Carolina
  - The Ohio State University, Columbus, Ohio
  - UPMC McKeesport, McKeesport, Pennsylvania
  - Vanderbilt University Medical Center - Vanderbilt Wound Center, Nashville, Tennessee
  - Richard C. Galperin DPM PA, Dallas, Texas
  - HCA Healthcare Houston Medical Center, Houston, Texas
  - Futuro Clinical Trials, LLC, McAllen, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Galiano RD, Li RA, Lantis JC, Oropallo A, Ulloa J, Iafrati M, Lavery LA, O'Connell J, Nouvong A. The trial design of the concurrent optical and magnetic stimulation (COMS) therapy study for refractory diabetic foot ulcers (MAVERICKS): a multicenter, randomized, sham-controlled, double-blind investigational device exemption clinical study. Wounds. 2025 Aug;37(8):275-282. doi: 10.25270/wnds/25037. PMID 40931367